CLINICAL TRIAL: NCT01691261
Title: Phase 1, Open-label, Safety and Feasibility Study of Implantation of Pf-05206388 (human Embryonic Stem Cell Derived Retinal Pigment Epithelium (rpe) Living Tissue Equivalent) in Subjects with Acute Wet Age Related Macular Degeneration and Recent Rapid Vision Decline
Brief Title: A Study of Implantation of Retinal Pigment Epithelium in Subjects with Acute Wet Age Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DACL1010; 2011-005493-37 (EudraCT Number)
Record Dates: First submitted 2012-09-19; First posted 2012-09-24 (Estimated); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): PF-05206388 Retinal Pigment Epithelium living tissue equivalent for intraocular use in the form of a monolayer of Retinal Pigmented Epithelial (RPE) cells immobilized on a polyester membrane
  Interventions: Biological: PF-05206388

INTERVENTIONS:
Biological: PF-05206388 — PF-05206388 will be provided as a Retinal Pigment Epithelium living tissue equivalent for intraocular use in the form of a monolayer of Retinal Pigmented Epithelial (RPE) cells immobilized on a polyester membrane. The membrane is approximately 6 mm x 3 mm and will contain a confluent layer of RPE cells, at a nominal dose of 17 mm2. The implant is intended to be life-long.

SUMMARY:
Phase 1 trial of retinal pigment epithelium replacement in subjects with wet age-related macular degeneration in whom there is rapidly progressing vision loss

DETAILED DESCRIPTION:
Phase 1, open-label, safety and feasibility study of implantation of PF-05206388 (human embryonic stem cell derived retinal pigment epithelium) in subjects with wet age related macular degeneration and rapid vision loss

ELIGIBILITY:
Inclusion Criteria:

* Male and /or post-menopausal female subjects aged 60 years or above.
* Diagnosis of wet Age-related Macular Degeneration (AMD) plus rapid recent vision decline
* An informed consent document signed and dated by the subject or a legal representative.

Exclusion Criteria:

* Pregnant females; breastfeeding females; and females of childbearing potential.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement, whichever is longer) or 5 half-lives preceding the first dose of study medication.
* Current or previous significant other ocular disease in the study eye, as determined by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events. | 52 weeks
  The number of Adverse Events (AE) and Serious Adverse Events (SAE) noted during the study and an assessment of whether they are trial product related
Change in baseline in ETDRS best corrected visual acuity (BCVA) - Proportion of subjects with an improvement of 15 letters or more at Week 24. | 24 weeks
  The number of patients with a difference between the baseline BCVA and BCVA at 24 weeks in ETDRS letters, where the differences is 15 letters or more, as a percentage of the total number of cases.

SECONDARY OUTCOMES:
Change in baseline in ETDRS best corrected visual acuity (BCVA) - Proportion of subjects with an improvement of 15 letters or more | Weeks 1,2,4,8, 12,16, 36, 52
  The number of patients with a difference between the baseline BCVA and BCVA at weeks 1,2,4,8, 12,16, 36, 52 in ETDRS letters, where the differences is 15 letters or more, as a percentage of the total number of cases.
Mean change of best corrected visual acuity (BCVA) from baseline by study visit. | 52 weeks
  The mean difference between the baseline BCVA and final BCVA in ETDRS letters for all cases
Position of PF-05206388 by serial biomicroscopic evaluation. | Day 2 and Weeks 1, 2, 4, 8, 10, 12, 16, 24, 36, 52
  Measurement of movement in millimetre and rotation in degrees measure relative to baseline, at day 2 and weeks 1, 2, 4, 8, 10, 12, 16, 24, 36 and 52
Position and presence of pigmented RPE cells by serial fundus photography | Weeks 2, 4, 8, 10, 12, 16, 24, 36, 52
  The subjective reporting of area of pigmentation as a % with cross reference to the OCT at weeks 2, 4, 8, 10, 12, 16, 24, 36 and 52
Mean change from baseline in contrast sensitivity by Pelli Robson test | Weeks 24, 52
  The mean difference between the baseline BCVA and final BCVA in Pelli Robson letters read, across all subjects
Change in liver and renal function by blood tests and liver ultrasound . | Weeks 24 and 52
  Record of any abnormalities in liver and renal function on blood testing and any abnormalities detected on the liver ultrasound.
Change in leakage or perfusion in normal fundal vasculature and presence of abnormal vasculature by fundus fluorescein angiography. | Weeks 4, 8, 12, 24 and 52
  Assessment and noting of abnormalities on Funded fluorescine angiography at weeks 4, 8, 12, 24 and 52.
Change in central 30 degree of visual function by Humphrey Field test. | Weeks 4, 8, 12, 24 and 52
  Recording and reporting of any changes on the central 30 degree field on the automated Humphrey Field test at weeks 4, 8, 12, 24 and 52
Change in thickness of RPE layer by B-mode orbital ultrasound. | Weeks 4, 8, 16, 24, 36, 52
  Recording of any changes in thickness of RPE layer by B-mode orbital ultrasound carried out by the ocular oncologist or medical physicist at weeks 4, 8, 16, 24, 36, 52.

CONTACTS AND LOCATIONS:
Overall Officials: Moorfields, Study Director — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4711001&StudyName=A%20Study%20Of%20Implantation%20Of%20Human%20Embryonic%20Stem%20Cell%20Derived%20Retinal%20Pigment%20Epithelium%20In%20Subjects%20With%20Acute%20Wet%20Age%20Related%20Macular